CLINICAL TRIAL: NCT03265041
Title: Predictors of Long Term Graft Patency After Coronary Artery Bypass Graft Surgery (Multi-slice CT Coronary Angiography Study Validated by Coronary Angiography)
Brief Title: Long Term Predictors of Graft Patency After Coronary Artery Bypass Graft Surgery (Multi-slice CT Coronary Angiography Study Validated by Coronary Angiography)
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Abdallah Hasaballah Farag, resident, Assiut University
Other Study IDs: CT coronary post CABG
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: multi-slice CT coronary angiography and coronary angiography — multi-slice CT coronary angiography to evaluate graft number and patency validated by coronary angiography

SUMMARY:
To detect and evaluate the predictors of graft patency after coronary artery bypass graft surgery as assessed by multi-slice CT coronary angiography validated by coronary angiography

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is an effective treatment of complex, multi-vessel coronary artery disease(1) .The majority of these patients receive left internal mammary artery (IMA) grafts to the left anterior descending (LAD) coronary artery and saphenous vein grafts (SVGs) or other conduits to the remaining vessels. Based on small studies of selected groups of patients, it is generally believed that SVGs have a 40% to 50% 10-year patency and that the LIMA has a 90% to 95% 10-year patency The success of coronary artery bypass grafting (CABG) is dependent on the long-term patency of the arterial and venous grafts.(2) Graft failure is a surrogate marker for future cardiac events, including repeat revascularization, myocardial infarction ,and death(3)(4). Vein graft occlusion in the perioperative period is due to thrombosis resulting from technical problems. Vein graft occlusion within the first year is attributed to intimal proliferation, although after 1 year, atherosclerosis is thought to be the dominant factor (5) . LIMA graft failure was defined as diffuse and >95% conduit narrowing ("string sign" When IMA graft failure occurs, technical error is the most common cause in the early postoperative period, while late (and rare) IMA failure include progressive fibro-intimal proliferation and atherosclerosis either in the IMA graft or in the native LAD vessel)(6) Traditionally, graft patency has been evaluated with coronary angiography (ICA) but, since the advent of multi-detector computed tomography (MDCT), the temptation to use a noninvasive and widely available technique to study coronary artery bypass graft (CABG) patients has been stronger. The introduction of scanners like 64-slice and 128-slice upwards-along with new scan protocols opens new perspectives in non-invasive assessment of graft patency.(7) The pooled sensitivity and specificity of detecting complete graft occlusions - according to( Barbero et al ,2016) ,was 99% and 99% respectively as compared to the standard of coronary angiography. (8) Computed tomographic angiography, labeled as Appropriate test for evaluation of bypass grafts and coronary anatomy (9)

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent coronary artery bypass graft surgery more than one year ago complaining of chest pain are included in the study from September 2017 to September 2018
* Written consent, free and informed

Exclusion Criteria:

* • Renal insufficiency (serum creatinine >1.6 mg/dl).

  * Contrast hypersensitivity.
  * Irregular heart rhythm (e.g. Atrial fibrillation).
  * Inability to hold breath for at least 10 seconds

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • All patients underwent coronary artery bypass graft surgery more than one year ago complaining of chest pain presented to Assuit university heart center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
detection of predictors of long term graft patency following CABG | 1 year
  a. Primary (main): evaluation of long term predictors of graft patency following coronary artery bypass graft surgery
  1. Clinical risk factors e.g Age, gender, smoking, Diabetus mellitus, hypertension, Dyslipidemia, chronic kidney disease, congestive heart failure, medications especially antiplatelet and statin therapy, beta-blockers and calcium channel blockers .
  2. Biochemical risk factors e.g HDL, LDL, Total cholesterol level
  3. Angiographic risk factors : competitive flow and degree of stenosis in the native vessels.

SECONDARY OUTCOMES:
Assessment of re-hospitalization rate following CABG | 1 year
Relation between type of the graft and graft patency | 1 year
Detection of sensitivity and specificity of CT coronary angiography for detection and assessment of graft patency | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Harskamp RE, Alexander JH, Ferguson TB Jr, Hager R, Mack MJ, Englum B, Wojdyla D, Schulte PJ, Kouchoukos NT, de Winter RJ, Gibson CM, Peterson ED, Harrington RA, Smith PK, Lopes RD. Frequency and Predictors of Internal Mammary Artery Graft Failure and Subsequent Clinical Outcomes: Insights From the Project of Ex-vivo Vein Graft Engineering via Transfection (PREVENT) IV Trial. Circulation. 2016 Jan 12;133(2):131-8. doi: 10.1161/CIRCULATIONAHA.115.015549. Epub 2015 Dec 8. PMID 26647082
- [Background] Di Lazzaro D, Crusco F. CT angio for the evaluation of graft patency. J Thorac Dis. 2017 Apr;9(Suppl 4):S283-S288. doi: 10.21037/jtd.2017.03.111. PMID 28540071
- [Background] Barbero U, Iannaccone M, d'Ascenzo F, Barbero C, Mohamed A, Annone U, Benedetto S, Celentani D, Gagliardi M, Moretti C, Gaita F. 64 slice-coronary computed tomography sensitivity and specificity in the evaluation of coronary artery bypass graft stenosis: A meta-analysis. Int J Cardiol. 2016 Aug 1;216:52-7. doi: 10.1016/j.ijcard.2016.04.156. Epub 2016 Apr 22. PMID 27140337
- [Background] TTE/TEE Appropriateness Criteria Writing Group; Douglas PS, Khandheria B, Stainback RF, Weissman NJ; TTE/TEE Appropriateness Criteria Technical Panel; Brindis RG, Patel MR, Alpert JS, Fitzgerald D, Heidenreich P, Martin ET, Messer JV, Miller AB, Picard MH, Raggi P, Reed KD, Rumsfeld JS, Steimle AE, Tonkovic R, Vijayaraghavan K, Yeon SB; ACCF Appropriateness Criteria Working Group; Hendel RC, Peterson E, Wolk MJ, Allen JM; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American Society of Echocardiography; American College of Emergency Physicians; American Society of Nuclear Cardiology; Society for Cardiovascular Angiography and Interventions; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance. ACCF/ASE/ACEP/ASNC/SCAI/SCCT/SCMR 2007 appropriateness criteria for transthoracic and transesophageal echocardiography: a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group, American Society of Echocardiography, American College of Emergency Physicians, American Society of Nuclear Cardiology, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, and the Society for Cardiovascular Magnetic Resonance. Endorsed by the American College of Chest Physicians and the Society of Critical Care Medicine. J Am Soc Echocardiogr. 2007 Jul;20(7):787-805. doi: 10.1016/j.echo.2007.06.011. No abstract available. PMID 17617305
- [Background] Goldman S, Zadina K, Krasnicka B, Moritz T, Sethi G, Copeland J, Ovitt T, Henderson W. Predictors of graft patency 3 years after coronary artery bypass graft surgery. Department of Veterans Affairs Cooperative Study Group No. 297. J Am Coll Cardiol. 1997 Jun;29(7):1563-8. doi: 10.1016/s0735-1097(97)82539-9. PMID 9180120
- [Background] Greenland P, Knoll MD, Stamler J, Neaton JD, Dyer AR, Garside DB, Wilson PW. Major risk factors as antecedents of fatal and nonfatal coronary heart disease events. JAMA. 2003 Aug 20;290(7):891-7. doi: 10.1001/jama.290.7.891. PMID 12928465